CLINICAL TRIAL: NCT05478317
Title: Esthetic Crown Lengthening With Closed Piezoelectric in Comparison to Open Flap Approach
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Augusta University (Other)
Responsible Party: Principal Investigator, Ahmed El-Awady, Assistant Professor, Augusta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1807704
Record Dates: First submitted 2022-07-19; First posted 2022-07-28 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Altered Passive Eruption of Teeth
Keywords: Crown lengthening; Open-flap approach; Piezoelectric approach

STUDY DESIGN:
Intervention Model Description: Subjects' matching inclusion criteria will be randomly assigned to control (OF) or tested (PZ) groups. After eligibility has been ascertained and consent has been obtained, subjects planned for ECL will be enrolled in the study and assigned to the group in 1:1 ratio using computer-generated block randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Crown lengthening using a traditional open-flap approach (OF). (Active Comparator): Esthetic Crown lengthening done using a traditional open-flap approach (OF).
  Interventions: Procedure: ECL-OF
- Test group: Crown lengthening using a minimally invasive approach by piezoelectric (PZ). (Experimental): Esthetic Crown lengthening done using a minimally invasive approach using piezoelectric (PZ).
  Interventions: Procedure: ECL- mPZ

INTERVENTIONS:
Procedure: ECL- mPZ — Flapless Technique using Piezoelectric (PZ):
  Gingivectomy and intra-sulcular incision will be carried out to remove strip of outlined marginal gingiva. However, no flap will be reflected the osseous recontouring will be carried using special piezoelectric tip below gingival margin. The required distance between the bone crest and the gingival margin will be checked by inserting a periodontal probe into the incision below gingival margin.
  Arms: Test group: Crown lengthening using a minimally invasive approach by piezoelectric (PZ).
Procedure: ECL-OF — Open Flap Technique (OF):
  Gingivectomy and intra-sulcular incision will be carried out to remove strip of outlined marginal gingiva. Full mucoperiosteal flap will be elevated to preform ostectomy and/or osteoplasty until the desired distance achieved between the bone crest and the gingival margin. After achieving the new supracrestal distance, the flap will be sutured.
  Arms: Control group: Crown lengthening using a traditional open-flap approach (OF).

SUMMARY:
In this randomized clinical trial, the investigators are comparing two different approaches for Esthetic crown lengthening- a minimally invasive approach using piezoelectric (PZ) and a traditional open flap approach (OF).

DETAILED DESCRIPTION:
The altered passive eruption is diagnosed when there is an excessive gingival display with short clinical crowns. Esthetic crown lengthening (ECL) is the most common surgical treatment of altered passive eruption. Traditional ECL involves osseous resection with gingivectomy or apical displaced gingiva. The amount of soft and hard tissue removal in this technique aims to provide a healthy and esthetically acceptable crown height. However, gingival tissue coronal rebound is one of the most noted post-operative complications of traditionally used techniques. On the other hand, surgical techniques that include flap reflection may cause more coronal displacement of the gingival margin. Hence, it is crucial to assess different surgical techniques to determine the most effective technique that gives the required outcomes with maximum patient satisfaction.

Piezoelectric bone surgery delivers high precision in resection, good tactile sensibility, and permits a selective cut of mineralized tissue while sparing soft tissue. Further, the minimally invasive technique (mECL) was suggested to reduce pain, post-op discomfort, and procedure duration, and to accelerate the healing process. The mECL technique conveys a potential alternative approach as a sutureless, atraumatic, and less invasive technique that has been shown to increase patient satisfaction and comfort. In addition, using piezoelectric for osseous resection in this closed approach increases the favorable surgical outcomes. However, the osseous resection in mECL may be incomplete and results in a coronal rebound on the gingival contour. In addition, osseous resection in this approach is very technique sensitive to avoid root damage and uneven bone resection. A few studies and even a fewer clinical trials evaluated the clinical outcome of mECL using piezoelectric for osseous resection (PZ). Hence, in this randomized clinical trial, gingival margin and bone crest stability will be evaluated after a minimally invasive approach using piezoelectric (PZ) and a traditional open flap approach (OF).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a gummy smile due to APE (Type 1B) in two or more maxillary anterior teeth
* Patients with normal muscular efficiency of the upper lip
* Patients with no vertical skeletal defects

Exclusion Criteria:

* Patients with systemic condition that prevent periodontal surgery
* Patients who smoke
* Patients with previous periodontal surgery in the same area
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2025-01-18 (Estimated); Study Completion 2025-01-18 (Estimated)

PRIMARY OUTCOMES:
Change of supracrestal width (cementoenamel junction to alveolar crest CEJ-AC) | CBCT parameter will be evaluated before the surgery and at 12 month after the surgery.
  Change of the supracrestal width will be measured using cone beam computed tomography (CBCT).

SECONDARY OUTCOMES:
Change on Probing depth (PD) | PD will be evaluated prior to surgery and 6 and 12 month after surgery
  Change on Probing depth (PD)
Change on Bleeding on probing (BOP) | BOP will be evaluated prior to surgery and 6 and 12 month after surgery
  Change on Bleeding on probing (BOP)
Change clinical attachment level (CAL). | CAL will be evaluated prior to surgery and 6 and 12 month after surgery
  Change on clinical attachment level (CAL).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Awady, BDS, MS, PHD, Principal Investigator — Augusta University
Locations (1):
- Augusta University-Dental College of Georgia, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No